CLINICAL TRIAL: NCT03181698
Title: Differences in Voxel-based Morphometry of Different Brain Structures in Patients With Mood Disorder Bipolar Mania in Comparison to Morphometry of Nrmal Controls
Brief Title: Brain Voxel-based Morphometry in Bipolar Mania
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaza Ragab, principal investigator, Assiut University
Other Study IDs: VBM MANIA
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Brain Voxel-based Morphometry in Mania
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- first group: patients with more than one episodes of mania
  Interventions: Diagnostic Test: Magnetic resonance imaging
- second group: sex-matched and age- matched healthy controls
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — A full Magnetic Resonance Imaging examination of the brain will be done for each of the subjects included in the study. The protocol of the study will include a high-resolution thin-cuts three Dimensions-T1 weighted gradient echo sequence to be used for the morphometric study.
  The obtained images will be analyzed for any gross structural abnormalities. by using fully-automated computational voxel-based volumetric software that calculates the volume of different structures of the brain. The obtained data will be analyzed statistically using linear regression tests to determine the differences between Bipolar Disorder type I mania patients and the healthy controls

SUMMARY:
Bipolar disorder is a complex psychiatric disorder characterized by recurrent episodes of mania or hypomania and depression, and affects around one to three percent of the population . Bipolar Disorder is associated with significant psychosocial morbidity and mortality , and is among the leading causes of disability worldwide . The disease is highly heritable, but the underlying pathophysiology is not yet understood .

DETAILED DESCRIPTION:
It is recognized that lesions in some specific neuro-anatomic areas due to brain disease, e.g., stroke or brain tumor, may lead to the development of secondary depression. The possibility of structural brain abnormalities as a cause of depression stimulated the use of structural brain imaging studies. Developments in structural neuroimaging by computed tomography and magnetic resonance imaging in the past 15 years facilitated the direct examination of specific brain structures, making the study of the relationship between anatomy and psychopathology is possible.

Neuro-anatomic model of mood regulation :

The prefrontal cortex has extensive connectivity to cortical and subcortical circuits that may underlie its importance in cognitive functions and modulation of limbic activity .The main subcortical structures participating in these circuits are the basal ganglia, thalamus, hypothalamus, brainstem, and the white matter tracts that connect these structures among themselves and to the cerebral cortex . A limbic-thalamic-cortical circuit consisting of the amygdala, the medio-dorsal nucleus of the thalamus, and the medial and ventro-lateral prefrontal cortex, and a limbic-striato-pallidal-thalamic circuit comprising the striatum, the ventral pallidum, and the components of the other circuit are the main neuro-anatomic circuits that have been proposed to participate in the pathophysiology of mood disorders.

The basal ganglia connect with cortical and limbic regions through circuits that, despite functioning segregated, are organized in parallel , in such a way that lesions in different parts of these circuits could result in malfunction. Additionally, the cerebellum, through connections with the brainstem and limbic structures, may also be involved in mood regulation.

Both primary and secondary mood disorders may involve abnormalities in specific fronto-subcortical neuro-anatomic circuits. Abnormalities in these brain regions or in contiguous areas that can affect the connections between these regions could reflect malfunction of these circuits, associated with development of mood disorders. Alternatively, abnormalities in these circuits could confer vulnerability to mood disorders, and its onset could be determined by interactions with environmental and genetic factors. Deficits during brain development due to these factors could result in under-development of particular brain areas, which could be related subsequently with mood disorders. The aging process or pathology such as vascular brain disease could result in atrophy of some of these regions. Thus, the influence of genetic, environmental, developmental, and degenerative factors during the development of these brain structures may determine the onset of mood disorders .

Although structural brain abnormalities in Bipolar Disorder have been reported, the pattern of structural brain abnormalities based on magnetic resonance imaging is still not clearly defined.

Aim of the study :

To study the morphometric criteria of different brain structures in patients with Bipolar Disorder type I mania in comparison to healthy subjects.

Subjects and Methods:

Patients :

Inclusion criteria:

Patients diagnosed to have mood disorder Bipolar I mania with or without psychotic features according to criteria of Diagnostic and statistical Manual of Mental disorder-IV (American Psychiatric Association 1994) by psychiatric sheath of psychiatric unit at Assiut University hospital .

The patients will be arranged in Two subgroups:

first group: twenty five patients in more than one episode second group: twenty age and sex-matched healthy subjects will be enrolled in the study

.

Exclusion Criteria:

first and second degree relatives of psychiatric patients will be excluded from the healthy controls.

Persons with any neurological disorder or other psychiatric illness will be excluded from controls Patients with proven major structural abnormality as detected during Magnetic resonance Imaging Examination will be excluded from patients or healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed to have mood disorder Bipolar I mania with or without psychotic features according to criteria of Diagnostic and Statistical Manual of Mental disorders-IV by psychiatric sheath of psychiatric unit at Assiut University hospital .

Exclusion Criteria:

1. first and second degree relatives of psychiatric patients will be excluded from the healthy controls.
2. Persons with any neurological disorder or other psychiatric illness will be excluded from controls
3. Patients with proven major structural abnormality as detected during Magnetic Resonance Imaging examination will be excluded from patients or healthy controls.

   -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed to have mood disorder Bipolar I mania with or without psychotic features according to criteria of Diagnostic and Statistical Manual of Mental disorders-IV by psychiatric sheath of psychiatric unit at Assiut University hospital .
  and sex and age-matched healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
mean differences in measurements of different brain structures | 2 hours
  mean differences in measurements of brain structures between patients of Mania and Healthy controls by using standard of all statistical parametric brain mapping-based processing software.voxels typically represent a volume of 27 mm3 (a cube with 3mm length sides)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hibar DP, Westlye LT, van Erp TG, Rasmussen J, Leonardo CD, Faskowitz J, Haukvik UK, Hartberg CB, Doan NT, Agartz I, Dale AM, Gruber O, Kramer B, Trost S, Liberg B, Abe C, Ekman CJ, Ingvar M, Landen M, Fears SC, Freimer NB, Bearden CE; Costa Rica/Colombia Consortium for Genetic Investigation of Bipolar Endophenotypes; Sprooten E, Glahn DC, Pearlson GD, Emsell L, Kenney J, Scanlon C, McDonald C, Cannon DM, Almeida J, Versace A, Caseras X, Lawrence NS, Phillips ML, Dima D, Delvecchio G, Frangou S, Satterthwaite TD, Wolf D, Houenou J, Henry C, Malt UF, Boen E, Elvsashagen T, Young AH, Lloyd AJ, Goodwin GM, Mackay CE, Bourne C, Bilderbeck A, Abramovic L, Boks MP, van Haren NE, Ophoff RA, Kahn RS, Bauer M, Pfennig A, Alda M, Hajek T, Mwangi B, Soares JC, Nickson T, Dimitrova R, Sussmann JE, Hagenaars S, Whalley HC, McIntosh AM, Thompson PM, Andreassen OA. Subcortical volumetric abnormalities in bipolar disorder. Mol Psychiatry. 2016 Dec;21(12):1710-1716. doi: 10.1038/mp.2015.227. Epub 2016 Feb 9. PMID 26857596
- [Background] Angst F, Stassen HH, Clayton PJ, Angst J. Mortality of patients with mood disorders: follow-up over 34-38 years. J Affect Disord. 2002 Apr;68(2-3):167-81. doi: 10.1016/s0165-0327(01)00377-9. PMID 12063145
- [Background] Tondo L, Isacsson G, Baldessarini R. Suicidal behaviour in bipolar disorder: risk and prevention. CNS Drugs. 2003;17(7):491-511. doi: 10.2165/00023210-200317070-00003. PMID 12751919
- [Background] Rocha-Rego V, Jogia J, Marquand AF, Mourao-Miranda J, Simmons A, Frangou S. Examination of the predictive value of structural magnetic resonance scans in bipolar disorder: a pattern classification approach. Psychol Med. 2014 Feb;44(3):519-32. doi: 10.1017/S0033291713001013. Epub 2013 Jun 5. PMID 23734914
- [Background] Soares JC, Mann JJ. The anatomy of mood disorders--review of structural neuroimaging studies. Biol Psychiatry. 1997 Jan 1;41(1):86-106. doi: 10.1016/s0006-3223(96)00006-6. PMID 8988799
- [Background] Lipska BK, Jaskiw GE, Weinberger DR. Postpubertal emergence of hyperresponsiveness to stress and to amphetamine after neonatal excitotoxic hippocampal damage: a potential animal model of schizophrenia. Neuropsychopharmacology. 1993 Aug;9(1):67-75. doi: 10.1038/npp.1993.44. PMID 8397725
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401